CLINICAL TRIAL: NCT07221786
Title: A Pilot Study of the Feasibility of Preoperative Opioid Tapering Before Spine Surgery Using Cognitive Behavioral Therapy and Measuring Postoperative Outcomes
Brief Title: Preoperative Opioid Tapering Before Spine Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Eric Schwenk, Professor of Anesthesiology and Perioperative Medicine, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB Control #22D.843_JT#25484
Record Dates: First submitted 2025-10-23; First posted 2025-10-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Opioid Consumption, Postoperative; Pain After Surgery; Opioid Dependency
Keywords: spine surgery; pain management; opioids; opioid use; depression; anxiety; opioid dependence; opioid tapering; cognitive behavioral therapy
MeSH Terms: conditions — Agnosia; Depression; Anxiety Disorders; Opioid-Related Disorders | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid tapering with Cognitive Behavioral Therapy (CBT) and education (Active Comparator): The CBT group will receive two preoperative sessions and at least one postoperative session conducted via telemedicine and performed by a pain psychologist. CBT sessions will focus on training in non-pharmacologic pain-coping skills, reducing the frequency and impact of negative pain-related cognitions and emotions, and on setting realistic behavioral goals.
  Patients will participate in the creation of an opioid tapering plan and will receive opioid education as well as education on how to taper opioids, the possibility of increased pain, the possibility of withdrawal symptoms, and the risks related to opioids, as well as the data on worsened perioperative outcomes in patients taking opioids.
  Interventions: Other: Opioid tapering with CBT and education
- Opioid tapering with education alone (Active Comparator): In this group patients will participate in the creation of an opioid tapering plan and will receive opioid education as well as education on how to taper opioids, the possibility of increased pain, the possibility of withdrawal symptoms, and the risks related to opioids, as well as the data on worsened perioperative outcomes in patients taking opioids.
  Interventions: Other: Opioid tapering with education alone

INTERVENTIONS:
Other: Opioid tapering with CBT and education — Patients in the opioid tapering plus CBT group will set up an initial meeting with the pain physician within a few days of enrollment to set the tapering schedule. They will also have two CBT appointments set up to complete via telemedicine during the time between enrollment and surgery.
  Arms: Opioid tapering with Cognitive Behavioral Therapy (CBT) and education
Other: Opioid tapering with education alone — Patients in this group will be instructed to continue their opioids at the same doses and frequencies they were taking up through the day of surgery. They will set up an initial meeting within a few days of enrollment with the chronic pain physician to determine the tapering schedule which will occur over 4 weeks or more leading into surgery. The patient and pain physician will collectively agree on a tapering schedule.
  Arms: Opioid tapering with education alone

SUMMARY:
This is a pilot study in which patients taking opioids chronically who are scheduled for spine surgery at least 4 weeks in advance will be randomly assigned to one of two groups: opioid tapering with education alone or opioid tapering with education plus cognitive behavioral therapy (CBT). The primary objective is to determine the proportion of each group that is successful in achieving their opioid tapering goals by the time of surgery.

DETAILED DESCRIPTION:
The perioperative period represents a particularly problematic time for opioid-dependent patients. Perioperative pain is often difficult to control, with opioid tolerance, opioid-induced hyperalgesia, and withdrawal making management a challenge. In addition to these short-term challenges, opioid-dependent patients experience poorer outcomes after surgery, including both early and late complications, emergency room visits, infections, and reoperations. Spine surgery in opioid-tolerant patients increases the risk for prolonged postoperative opioid use. This risk is in addition to the risk of prolonged opioid use that surgery itself introduces. The high prevalence of opioid use in spine patients makes spine surgery an ideal surgical model in which to study opioid tapering.

This is a randomized, controlled pilot study of 45 opioid-dependent patients undergoing spine surgery. Patients will be assigned in parallel to one of the following: 1. opioid tapering with education alone or 2. opioid tapering with education plus cognitive behavioral therapy (CBT). While all patients will meet with a pain physician to design a personalized tapering program, the CBT group will receive two CBT sessions prior to surgery. Pain, depression, anxiety, and opioid withdrawal will be assessed throughout the month prior to surgery and managed appropriately. Opioid use at the time of surgery will be assessed along with pain and depression and anxiety. Hospital outcomes, including pain, opioid use, quality of recovery, and postoperative complications, will be measured. Patients will be followed upon discharge by a chronic pain physician and patients assigned to CBT will receive one additional session after surgery. All patients will also be assessed via telephone call or Zoom at 30, 90, 180, and 365 days for pain, function, and opioid use.

ELIGIBILITY:
Inclusion:

* at least 18 years old
* scheduled for major spine surgery (i.e. at least 2 levels of fusion) with hospital admission of at least one night
* scheduled for spine surgery at least 4 weeks ahead of time
* takes between 40 and 200 oral morphine equivalents daily

Exclusion:

* inability to use a computer or tablet for telemedicine encounters
* non-English-speaking
* inability to complete assessments
* positive screen on the Columbia Suicide Screening Assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
proportion that achieved opioid tapering goal | Perioperative prior to surgery (postoperative day 0)
  Achievement of the opioid tapering goal for each patient will be assessed on day of surgery and will be based on average daily OMEs taken during the three days before surgery. The opioid tapering goal will be made on the initial visit with the study pain physician and will be specific to each patient.

SECONDARY OUTCOMES:
Brief Pain Inventory | Baseline, weeks 1-4 before surgery, day of surgery (postoperative day 0), postoperative days 1-3, and postoperative days 30, 90, 180 and 365.
  Brief Pain Inventory is a validated pain assessment tool that measures pain severity and its effects on daily function.
Clinical Opiate Withdrawal Scale | Baseline, once weekly on weeks 1-4 prior to surgery, day of surgery (postoperative day 0), postoperative day 1, and postoperative days 30, 90, 180, and 365.
  Standardized assessment of opioid withdrawal
Patient Health Questionnaire-9 | Baseline, weeks 1-4 prior to surgery, and postoperative days 30, 90, 180, and 365
  Depression screening
Generalized Anxiety Disorder-2 | Baseline
  Standardized generalized anxiety screening
Columbia Suicide Screening Assessment | Screening period
  This is a suicide risk screening tool
Daily opioid use in hospital | Postoperative days 0-7
  This will be the average daily opioid use in the hospital
Hospital length of stay | Postoperative days 0-7
  Duration of hospital stay in days
Quality of recovery-15 | Preoperative baseline, postoperative days 1-2
  This is a validated 15-question assessment of quality of recovery
Hospital Anxiety and Depression Scale | Postoperative days 0-3
  Anxiety and depression assessment for the hospitalization
Opioid use in daily OMEs | Day of surgery (postoperative day 0), postoperative days 30, 90, 180 and 365
  Patient-reported daily opioid use on average in mg
Daily opioid use in OMEs from prescription drug monitoring program | Day of surgery (postoperative day 0), postoperative days 30, 90, 180, and 365
  This is the prescribed daily opioids confirmed from the PDMP.
Nausea and vomiting | Postoperative days 0, 1, 2, 3, 30, 90, 180, and 365
  Nausea and vomiting measured on the following scale: 0=AE not experienced; 1=AE experienced but no treatment needed; 2=AE experienced and treatment was effective; 3=AE experienced and treatment was ineffective
Constipation | Postoperative days 0, 1, 2, 3, 30, 90, 180, and 365
  Constipation: 0=AE not experienced; 1=AE experienced but no treatment needed; 2=AE experienced and treatment was effective; 3=AE experienced and treatment was ineffective
Pruritus | Postoperative days 0, 1, 2, 3, 30, 90, 180, and 365
  Puritus: 0=AE not experienced; 1=AE experienced but no treatment needed; 2=AE experienced and treatment was effective; 3=AE experienced and treatment was ineffective
Patient satisfaction with pain control | Postoperative days 0, 1, 2, 3, 30, 90, 180, and 365
  0-10 scale with 0 being worst possible pain control and 10 being best possible pain control
SF-12 | Baseline, day of surgery (postoperative day 0), and postoperative days 30, 90, 180, and 365
  This is a brief assessment of physical and mental function

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadephia, Pennsylvania, United States

REFERENCES:
- [Background] Darnall BD, Roy A, Chen AL, Ziadni MS, Keane RT, You DS, Slater K, Poupore-King H, Mackey I, Kao MC, Cook KF, Lorig K, Zhang D, Hong J, Tian L, Mackey SC. Comparison of a Single-Session Pain Management Skills Intervention With a Single-Session Health Education Intervention and 8 Sessions of Cognitive Behavioral Therapy in Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Netw Open. 2021 Aug 2;4(8):e2113401. doi: 10.1001/jamanetworkopen.2021.13401. Erratum In: JAMA Netw Open. 2022 Apr 1;5(4):e229739. doi: 10.1001/jamanetworkopen.2022.9739. PMID 34398206
- [Background] Hassamal S, Haglund M, Wittnebel K, Danovitch I. A preoperative interdisciplinary biopsychosocial opioid reduction program in patients on chronic opioid analgesia prior to spine surgery: A preliminary report and case series. Scand J Pain. 2016 Oct;13:27-31. doi: 10.1016/j.sjpain.2016.06.007. Epub 2016 Jul 4. PMID 28850531
- [Background] Bicket MC, Gunaseelan V, Lagisetty P, Fernandez AC, Bohnert A, Assenmacher E, Sequeira M, Englesbe MJ, Brummett CM, Waljee JF. Association of opioid exposure before surgery with opioid consumption after surgery. Reg Anesth Pain Med. 2022 Jun;47(6):346-352. doi: 10.1136/rapm-2021-103388. Epub 2022 Mar 3. PMID 35241626
- [Background] Kalakoti P, Volkmar AJ, Bedard NA, Eisenberg JM, Hendrickson NR, Pugely AJ. Preoperative Chronic Opioid Therapy Negatively Impacts Long-term Outcomes Following Cervical Fusion Surgery. Spine (Phila Pa 1976). 2019 Sep;44(18):1279-1286. doi: 10.1097/BRS.0000000000003064. PMID 30973507
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Sun EC, Darnall BD, Baker LC, Mackey S. Incidence of and Risk Factors for Chronic Opioid Use Among Opioid-Naive Patients in the Postoperative Period. JAMA Intern Med. 2016 Sep 1;176(9):1286-93. doi: 10.1001/jamainternmed.2016.3298. PMID 27400458
- [Background] Reyes AA, Canseco JA, Mangan JJ, Divi SN, Goyal DKC, Bowles DR, Patel PD, Salmons HI, Morgenstern M, Anderson DG, Rihn JA, Kurd MF, Hilibrand AS, Kepler CK, Vaccaro AR, Schroeder GD. Risk Factors for Prolonged Opioid Use and Effects of Opioid Tolerance on Clinical Outcomes After Anterior Cervical Discectomy and Fusion Surgery. Spine (Phila Pa 1976). 2020 Jul 15;45(14):968-975. doi: 10.1097/BRS.0000000000003511. PMID 32604353
- [Background] Colvin LA, Bull F, Hales TG. Perioperative opioid analgesia-when is enough too much? A review of opioid-induced tolerance and hyperalgesia. Lancet. 2019 Apr 13;393(10180):1558-1568. doi: 10.1016/S0140-6736(19)30430-1. PMID 30983591